CLINICAL TRIAL: NCT00278616
Title: High Dose Cyclophosphamide & CAMPATH-1H With Hematopoietic Stem Cell Transplantation in Patients With Refractory Antiphospholipid Syndrome (APS): A Phase I Trial
Brief Title: Hematopoietic Stem Cell Transplantation in Patients With Antiphospholipid Syndrome
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU APS AUTO 2004
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: ANTIPHOSPHOLIPID SYNDROME
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Stem Cell Transplantation — Autologous Stem Cell Transplantation

SUMMARY:
Antiphospholipid syndrome is disease believed to be due to immune cells, cells which normally protect the body, but are now producing the protein which leads to abnormal clotting in the body. This study is designed to examine whether treating patients with high dose cyclophosphamide together with CAMPATH (drugs which reduce the function of the immune system), followed by return of the previously collected stem cells will result in improvement in the disease. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the intense chemotherapy is to destroy the cells in the immune system which may be causing the disease. The purpose of the stem cell infusion is to produce a normal immune system that will no longer attack the body. The study purpose is to examine whether this treatment will result in improvement in the disease. The drugs used in this study treatment are drugs for commonly used for immune suppression.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years< 55 years at the time of pretransplant evaluation
2. A or 6.12.B:

A) An established diagnosis of a definite primary APS by Sapporo criteria as follows:

1. Positive LA and/or ACLA IgG or IgM on two separate measurements, AND
2. Arterial, venous or small vessel thrombosis (confirmed by imaging or doppler studies or histopathology, with the exception of superficial venous thrombosis) OR pregnancy morbidity (defined as three or more embryonic losses, OR one or more premature birth due to preeclampsia or growth retardation, OR one or more fetal death)

B) APLA-positive Sneddon syndrome defined as an association of ischemic cerebrovascular events and a widespread livedo reticularis

3. Patients failed treatment with anticoagulation including warfarin, heparin/LMWH in the presence of positive LA and/or ACLA IgG, or IgM. Failure is defined as any of above described thromboembolic events (6.12.A-2 or 6.12.B) except for pregnancy morbidity while receiving therapeutic anticoagulation. Therapeutic anticoagulation is defined as at least 5000 U of regular heparin SQ BID, OR unfractionated IV heparin adjusted for therapeutic PTT, OR at least 40 mg of lovenox SQ QD (or equivalent LMWH), OR coumadin adjusted for INR of at least 2.0, documented within 1 month of a refractory event or within 3 months if patient was known to be previously stable PLUS in the opinion of the investigator the individual has been receiving adequate anticoagulation.

Exclusion Criteria:

1. Poor performance (PS) status (ECOG >2) at the time of entry, unless decline of PS is due to the disease itself and considered to be reversible.
2. Significant end organ damage such as (not caused by APS):

   * LVEF<40% or deterioration of LVEF during exercise test on MUGA or echocardiogram.

     * Untreated life-threatening arrhythmia.
     * Active ischemic heart disease or heart failure.
     * DLCO<40% or FEV1/FEV < 50%.
     * Serum creatinine >2.5 or creatinine clearance <30ml/min.
     * Liver cirrhosis, transaminases >3x of normal limits or bilirubin >2.0 unless due to Gilbert disease.

       3. HIV positive.

       4.Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.

       5. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.

       6. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.

       7. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.

       8. Inability to give informed consent.

       9. Major hematological abnormalities such as platelet count less than 100,000/ul, ANC less than 1000/ul unless due to APS.

       10. Failure to collect at least 2.0 x 106 CD34+ / kg cells.*

       11. Patients who are already in a clinical trial for APS treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Toxicity; Survival;Disease improvement;Time to disease progression; | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Background] Statkute L, Traynor A, Oyama Y, Yaung K, Verda L, Krosnjar N, Burt RK. Antiphospholipid syndrome in patients with systemic lupus erythematosus treated by autologous hematopoietic stem cell transplantation. Blood. 2005 Oct 15;106(8):2700-9. doi: 10.1182/blood-2005-01-0330. Epub 2005 May 3. PMID 15870182